CLINICAL TRIAL: NCT03573999
Title: Effect of Isosmotic Doses of Mannitol 20% Versus Hypertonic Saline 7.5% in Brain Metabolism and Oxygenation in Supratentorial Craniotomies
Brief Title: Effect of Mannitol 20% Versus Hypertonic Saline 7.5% in Brain Metabolism and Oxygenation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgia Tsaousi, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OsmoMetOx
Record Dates: First submitted 2018-05-20; First posted 2018-06-29 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2020-01

CONDITIONS: Brain Edema; Metabolic Disturbance; Electrolyte and Fluid Balance Conditions
Keywords: mannitol; hypertonic saline; brain metabolism; brain oxygenation
MeSH Terms: conditions — Brain Edema | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol 20% (Active Comparator): Mannitol 20% (4.6ml/kg) will be administered 20 minutes before dura matter opening.
  Interventions: Drug: Mannitol
- Hypertonic saline 7.5% (Experimental): Hypertonic saline 7.5% (2ml/kg) will be administered 20 minutes before dura matter opening
  Interventions: Drug: NaCl 7.5%

INTERVENTIONS:
Drug: Mannitol — 4.6 ml/kg will be administered before dura opening
  Arms: Mannitol 20%
Drug: NaCl 7.5% — 2 ml/kg will be administered before dura opening
  Arms: Hypertonic saline 7.5%

SUMMARY:
Usage of osmotic agents is a standard practice in neuroanesthesia since cerebral edema is a very common situation for patients with pathology in the brain. Cerebral edema is defined as the accumulation of fluid in the intracellular or extracellular compartments of the brain. Among other situations that have nothing to do with the brain, a supratentorial pathology such as a tumor, traumatic injury or an aneurysm, will lead to disruption of blood-brain barrier, and energy crisis of the cells that will cause mainly vasogenic and cytotoxic cerebral edema. The most common monitoring method for "measuring" cerebral edema is ICP (intracranial pressure) in which normal values are (with differences in the bibliography) 10-15 mmHg.

The osmotic agents used most in neuroanesthesia are mannitol 20% and hypertonic NaCl 7.5% or 3%. Their brain relaxation effectiveness is supposed to be quite the same between the two different agents. Their main difference is that mannitol induces diuresis. Also, electrolyte disorders are another possibility after mannitol infusion. On the other hand, NaCl 7.5% causes vasodilation, does not induce diuresis and hemodynamically, even though it reduces SBP, it raises CO because of its excessive vasodilation. But both reduce cerebral edema due to the change of osmotic pressure in the vessels, that leads to extracting water from brain cells.

A supratentorial craniotomy is de facto worsening the oxygenation and metabolism condition of the surgical site, adding to the problem the intracranial pathology causes in the first place. So if oxygen provided is low and the metabolic rate is high, the rate of anaerobic metabolism will raise. Measuring the oxygen in the jugular bulb is the most reliable monitoring method of cerebral oxygenation and metabolism.

It becomes evident that optimization of cerebral oxygenation during a craniotomy will possibly affect the outcome of a patient, by improving it. So, if any superiority of one osmotic agent over the other could be demonstrated this will be very helpful in the decision making in routine clinical practice.

DETAILED DESCRIPTION:
Each participant will receive standard monitoring (ECG, SpO2, SBP, BIS, urine output, temperature). More detailed hemodynamic monitoring will be obtained by Edwards Lifesciences ClearSight system (CO, CI, SV, SVI, SVV, SVR, SVRI).

TCI Propofol and Remifentanil will be the agents of choice for induction and maintenance in anesthesia and cisatracurium will be used for neuromuscular blockade for intubation.

Protective mechanical ventilation will be chosen (7ml/kg IBW) with a Respiratory rate to obtain a PaCO2 of 35-40 mmHg. PEEP will be changed for the best PaO2/FiO2 ratio and FiO2 of choice will be 0.5.

The radial artery catheterization will be applied for direct blood pressure measurement and arterial blood gas sampling ( pH, PaO2, PaCO2, HCO3, BE, Osmolality, Lactic acid, Hb, Glucose, Na, K will be measured).

The jugular bulb ipsilateral to the craniotomy site will be catheterized for receiving blood samples for blood gas analysis. The following oxygenation and metabolic parameters / derivates will be measured or calculated: SjvO2, pH, PjvO2, PjvCO2, HCO3, BE, Osmolality, Lactic acid jv, Hb, Glucose, Na, K, AjvDO2, AjvCO2, O2ERbr, eRQbr, AjvDL, and LOI.

The osmotic agent will be administered 20 minutes before dura matter incision. Before the dura mater opening the subdural space pressure will be measured and relevant CPP will be calculated. Brain Relaxation Score will be assessed by the neurosurgeon.

Phases

* T0: 5 minutes before administration of the osmotic agent
* T15: 15 minutes after administration of the osmotic agent
* T30: 30 minutes after administration of the osmotic agent
* T60: 60 minutes after administration of the osmotic agent
* T90: 90 minutes after administration of the osmotic agent
* T120: 120 minutes after administration of the osmotic agent
* T180: 180 minutes after administration of the osmotic agent
* T240: 240 minutes after administration of the osmotic agent Blood samples for measuring S-100b will be collected at phases T0, T240 and 12 hours after osmotic agent administration.

Postoperative complications, length of ICU stay, GOS-E (Glasgow Outcome Scale) and other neurological deficits will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 75 years
* ASA Physical status 1 to 3
* Elective or semi-elective supratentorial craniotomy
* Signed informed consent

Exclusion Criteria:

* Craniotomy for suprasellar pathologies
* Re-craniotomy at the same site
* Perioperative sodium disorders (Na <130 mEq/L or >150 mEq/L)
* Administration of intravenous mannitol or hypertonic saline 7.5% 24 hours or less before the surgery
* Preoperative obstructive hydrocephalus
* Congestive heart failure
* Renal failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Changes of jugular venous oxygen saturation | 15 minutes after the end of the infusion of the tested osmotic agent
  Alterations in jugular venous oxygen saturation (%) after intravenous infusion of isosmotic doses of mannitol 20% and hypertonic saline 7.5%

SECONDARY OUTCOMES:
Changes of S-100b protein | 6 hours after the end of the infusion of the tested osmotic agent
  Alterations in S-100b (μg/L) after intravenous infusion of isosmotic doses of mannitol 20% and hypertonic saline 7.5%
Changes in the cardiac index | 15 minutes after the end of the infusion of the tested osmotic agent
  Alterations in the cardiac index (L/min/m2) after intravenous infusion of isosmotic doses of mannitol 20% and hypertonic saline 7.5%
Brain tension after intravenous infusion of isosmotic doses of mannitol 20% and hypertonic saline 7.5% assessed by Brain relaxation Score and subdural pressure | 2 minutes before dura opening
  Brain tension graded from 1 to 4 (1 indicates satisfactory brain relaxation and 4 serious brain bulking)
Functional outcome of participants | 7 days post surgery
  Functional status of the participants assessed by Extended GOS ranginging from 1 to 7 (1 indicates death and 7 neurologically intact patient)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Tsaousi, Principal Investigator — Aristotle University Of Thessaloniki
Locations (2):
- Greece (2):
  - AHEPA University Hospital, Thessaloniki
  - Georgia Tsaousi, Thessaloniki

IPD SHARING:
Plan to Share IPD: No